CLINICAL TRIAL: NCT05171062
Title: Safety and Tolerability of Bexmarilimab Plus Pembrolizumab for Patients With Advanced (Inoperable or Metastatic) Non-small Cell Lung Cancer (NSCLC)
Brief Title: Dose Escalation Trial of Bexmarilimab (FP-1305) Plus Pembrolizumab in Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants were enrolled, the study was inactivated with the IRB on May 15, 2023. The sponsor notified the PI that a Phase II trial had been allowed to proceed by the FDA.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Faron Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 21-0153; 20210791HU (Other: UT Health San Antonio)
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — bexmarilimab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose levels will be escalated to determine maximum tolerated dose (MTD) in participants with non-small cell lung cancer (NSCLC) eligible for standard of care pembrolizumab treatment. MTD will be determined based on occurence of dose limiting toxicities (DLTs) by standard 3+3 escalation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Study patients will receive 0.1-1 mg/kg bexmarilimab (FP-1350) given in combination with Pembrolizumab 200mg IV once every three weeks. The first subject will be started on 0.1mg to establish toleration, for one dose, and then the dose will be escalated to 1mg. This subject will be included in Cohort 1 data.
  Interventions: Drug: bexmarilimab (FP-1305); Drug: Pembrolizumab
- Cohort 2 (Experimental): Study participants will receive 3mg/kg Bexmarilimab given in combination with Pembrolizumab 200mg IV once every three weeks. 3 participants will need to complete this level before the next cohort dosing begins.
  Interventions: Drug: bexmarilimab (FP-1305); Drug: Pembrolizumab
- Cohort 3 (Experimental): Study participants will receive 10 mg/kg Bexmarilimab plus pembrolizumab 200mg IV once every 3 weeks. 3 participants will need to complete this level before the next cohort dosing begins.
  Interventions: Drug: bexmarilimab (FP-1305); Drug: Pembrolizumab
- Cohort 4 (Experimental): Study participants will receive 30 mg/kg Bexmarilimab plus pembrolizumab 200mg IV once every 3 weeks.
  Interventions: Drug: bexmarilimab (FP-1305); Drug: Pembrolizumab

INTERVENTIONS:
Drug: bexmarilimab (FP-1305) — standard 3+3 dose escalation trial of bexmarilimab (FP-1305)
  Other Names: FP-1305
Drug: Pembrolizumab — Pembrolizumab 200mg IV is administered in 4 planned bexmarilimab dose escalation cohorts
  Other Names: Keytruda

SUMMARY:
This study enrolls patients with Non-small cell lung cancer and treats them with the investigational drug Bexmarilimab (FP-1305) plus standard of care Pembrolizumab to block Common lymphatic endothelial and vascular endothelial receptor-1 (CLEVER-1). Treating with an antiCLEVER-1 antibody, such as bexmarilimab, could lead to immune system activation, which, in turn, may lead to cancer elimination.

DETAILED DESCRIPTION:
This study is an open label, Phase Ib, standard 3+3 dose escalation trial of bexmarilimab (FP-1305) plus pembrolizumab in 4 planned dose escalation cohorts in Non-Small Cell Lung Cancer (NSCLC) to determine the safety and tolerability of repeated doses of bexmarilimab plus pembrolizumab administered in three-week intervals (Q3W) (Figures 1 and 2) defined as treatment cycles. Bexmarilimab is a monoclonal antibody to common lymphatic endothelial and vascular endothelial receptor-1 (CLEVER-1), administered by IV infusion every 3 weeks. Pembrolizumab is a monoclonal antibody to programmed death-1 (PD-1), administered by 30-minute IV infusion every 3 weeks. When pembrolizumab and bexmarilimab are given on the same day, bexmarilimab is given before pembrolizumab. No pre-medication(s) is/are needed before infusion of either drug.

Dose levels will be escalated to determine the maximum tolerated dose (MTD) in trial subjects with NSCLC eligible for pembrolizumab as standard of care (SOC) treatment. The MTD level will be determined based on the occurrence of dose limiting toxicities (DLTs) by standard 3+3 escalation. For the purposes of DLT, only DLT attributable to or likely due to bexmarilimab are counted. DLTs clearly related to pembrolizumab do not count as DLTs for the purposes of dose escalation. The pre-determined dose levels in the dose escalation part are 0.1, 1.0, 3.0, 10.0, and 30 mg/kg, In Cohort 0, if the first dose at 0.1 mg/kg is tolerated, that patient will advance to Cohort 1 to finish the trial at the Cohort 1 bexmarilimab dose. Dose escalation within individual patients beyond Cohort 0 is not permitted.

Beyond the Level 0 dose level, each subject will be observed for three weeks for DLT (subject at Level 0 will advance to the next level after a 3-week observation period). In the absence of DLT, once three subjects have received the second dose at dose level (for example at Level 1), each of them with a minimum of three-week follow-up, the dose is escalated to the third dose level (in this example to Level 2). If a subject is withdrawn/discontinued for any reason or dies before the completion of Cycle 3, week 1, the withdrawn/discontinued subject must be replaced with a new subject enrolled at the same dose level until three subjects have reached the three-week follow-up and the dose escalation to the next level may occur.

The dose cannot be escalated to the next level before a three-week DLT period is reached for all the subjects at the current level. Beyond Level 0, if subjects fail to reach the three-week DLT window in a given cohort for any reason, they must be replaced, and the replacement subject will be observed accordingly before escalation can proceed. If a subject misses a dose in the DLT period that subject must be replaced so that each subject receives 2 doses of bexmarilimab in the DLT window.

Once a DLT is observed in any of the treated patients, an additional 3 subjects will be enrolled at this dose. If no further DLTs are observed, escalation proceeds as planned. If a second DLT occurs, the MTD is defined as the prior cohort. A maximum of 36 evaluable subjects will be accrued for the MTD determination.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written Informed Consent
2. Aged ≥ 18 years
3. Tumor sample obtained less than six months from the date of consent
4. Histologically confirmed NSCLC eligible for pembrolizumab as standard of care
5. Known tumor PD-L1 TPS score
6. Measurable disease based on RECIST 1.1 as determined by the site
7. Women of child-bearing potential must have a negative pregnancy test prior to trial entry and cycle 1 day 1 and should not be breast feeding.
8. Women of child-bearing potential and men who have partners of child-bearing potential must be willing to practice highly effective contraception for the duration of the trial and for three months after the completion of treatment

Exclusion Criteria:

1. Less than 21 days since the last dose of intravenous anticancer chemotherapy or less than five half-lives from a small molecule targeted therapy or oral anticancer chemotherapy before the first bexmarilimab administration
2. Any immunotherapy within preceding 3 weeks from the first bexmarilimab administration
3. Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period. Subjects whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have returned to baseline or resolved. Any steroids administered as part of this therapy must be completed at least three days prior to study medication.
4. Investigational therapy or major surgery within 4 weeks from the date of consent
5. Active clinically serious infection >grade 2 NCI-CTCAE version 5.0 (Appendix 6) within preceding 2 weeks from the date of consent
6. Subject has not recovered from the previous therapies to Grade 1 severity as classified by the NCI-CTCAE version 5.0 (except Grade 2 alopecia, neuropathy or thyroid disorders)
7. Pregnant or lactating women
8. The subject requires systemic corticosteroid or other immunosuppressive treatment
9. Use of live (attenuated) vaccines for 30 days prior to the start of study treatment, d during treatment, and until last visit
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Subject is unwilling or unable to comply with treatment and trial instructions
12. Any condition that study investigators consider an impediment to safe trial participation
13. Prior therapy for advanced stage or metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Cycle 2 plus 3 weeks (21 days following the first dose of both study drugs)
  Measured by the number of adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse events (NCI-CTCAE v. 5) ≥Grade 3 occuring during the 21 days 3 weeks) following the first dose of bexmarilimab plus pembrolizumab in Cycle 2 and related to bexmarilimab are considered dose limiting toxicity (DLT) with the following exceptions:
  * Grade 3 infusion reactions that resolve within 8 hours from the onset of the reaction and are not defined as a DLT
  * For nausea/vomiting/diarrhea, only adequately pre-treated grade 3 or 4 toxicity will qualify as DLT
  * For thrombocytopenia, hemorrhage is required to qualify grade 3 toxicity as DLT; grade 4 thrombocytopenia is DLT regardless of hemorrhaged
  * For neutropenia, fever is required to qualify grade 3 toxicity as DLT. A duration > 5 days is required to qualify grade 4 toxicity as DLT
Programmed Death Cell Ligand 1 (PD-L1) level | Cycle 1 (21 days), pre-dose levels at start of Cycle 3 (42 days)
  Measured using analysis of soluble CLEVER-1 (sClever) levels

SECONDARY OUTCOMES:
Immunophenotyping | Baseline to study end (approximately 12 months)
  Assessed by measurement of the circulating immune cell populations in serum over time

OTHER OUTCOMES:
Objective Response Rate (ORR) | Cycle 1 (21 days)
  The reported proportion of subjects of all evaluable subjects within each tumor type cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Supreet Kaur, MD, Principal Investigator — UT Health San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided